CLINICAL TRIAL: NCT04558177
Title: Repetitive Transcranial Stimulation to Treat Depression and Anxiety in Senior Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Glenrose Foundation (Other); Centre for Aging and Brain Health Innovation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00078317
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Geriatric In-patients
Keywords: depression; anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: double blind placebo controlled
Who Masked: Participant, Care Provider
Masking Description: sham procedure appears indistinguishable from intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation Group (Experimental): Will receive ~1.5mA transcranial stimulation for 20 minutes, 5x per week from a direct current stimulator
  Interventions: Device: Direct current stimulator
- Device placed only, no stim (Sham Comparator): Same as experimental group but the stimulation from the direct current stimulator will be initiated and then stopped
  Interventions: Device: Direct current stimulator

INTERVENTIONS:
Device: Direct current stimulator — HDCprog connected to a direct current stimulator, controls the number of stimulations (maximum 99), the intensity (up to 1.5mA per channel), the duration (maximum 20min), and the minimum interval between two consecutive simulations (max 1168 hours). A sham condition is also available which will ramp the stimulation to a preset maximum level and then immediately reduces the stimulation to 0.

SUMMARY:
Many seniors admitted for rehabilitation have symptoms of depression and anxiety that need to be treated before they can effectively engage in rehabilitation therapy. Anti-depressant or anti-anxiety medications are often used but there are many reasons why alternative or adjunctive treatments may be desirable. Medications can take weeks to become effective, if they work at all. There are many potential side effects of medications, especially in an older population, including cognitive and other neurologic impairments. There is also an increasing resistance to a polypharmacy approach to treatment in this population. A low-risk, relatively non-invasive, easily applied and well-tolerated treatment to accelerate mood and anxiety disorder resolution would allow earlier and more effective engagement in rehabilitation therapy. This would in turn shorten lengths of stay and improve quality of life. Recently, trans-cranial direct current stimulation with 1-2 mA currents has been proposed as a potential innovative alternative treatment modality. This stimulation is safe, easy to use, relatively insensitive to electrode placement, and may have other beneficial cognitive effects. The stimulation device consists of two electrodes placed on either side of the head, a unit that provides the stimulation and wires that connect this unit to the electrodes will be used. The electrodes are held in place with a head band.

DETAILED DESCRIPTION:
Purpose: To determine if using adjunctive TDCS to treat seniors admitted with symptoms of depression and anxiety reduces length of stay and improves quality of life. Hypothesis: Using transcranial direct current stimulation (TDCS) will decrease length of stay because it will reduce symptoms of depression and anxiety enabling patients to engage with their therapy sooner and more effectively. Justification: Anti-depressant or anti-anxiety medications are often used for this inpatient population but there are many reasons why alternative or adjunctive treatments may be desirable. Medications can take weeks to become effective, if they work at all. There are many potential side effects of medications, especially in an older population, including cognitive and other neurologic impairments. There is also an increasing resistance to a polypharmacy approach to treatment in this population. A low-risk, relatively non-invasive, easily applied and well-tolerated treatment to accelerate mood and anxiety disorder resolution would allow earlier and more effective engagement in rehabilitation therapy. This would in turn shorten lengths of stay and improve quality of life. Objectives: to determine if (1) TDCS reduces symptoms of depression and anxiety and (2) if patients in the intervention group are discharged from hospital sooner than those in the sham group. Research Method/Procedure: Direct current of 1.5 milliamp (mA) will be applied for 20 minutes 5x/week for 3 weeks in a hemispheric montage over the homologous dorso-lateral prefrontal cortices, anodal on the left. The Glenrose Rehabilitation Hospital is Canada's largest freestanding rehabilitation institution with programs and services for all age groups. Rehabilitation services cover all disciplines from physical, occupational therapy to social work. Older adults are admitted to 3D and 4C to address issues related to frailty such as weakness and poor balance which affect ability to undertake activities of daily living. Most of the services they receive as inpatients come from physical and occupational therapists with speech therapists and psychologists also available if needed.Patients will be drawn from these seniors admitted to these 2 geriatrics units, 3D and 4C. Candidates who meet the eligibility criteria and are interested in the project will be approached by the RA who is not involved in their care and will seek their consent. Patients will be randomized into standard care (SoC) plus active TDCS and SoC with sham TDCS. TDCS is unique in that effective double blind sham conditions can be created. Effectiveness of treatment will be judged primarily on reduced length of stay with improved Geriatric Depression Score (GDS), Geriatric Anxiety Score (GAS) and Older Person's Quality of Life (OPQOL) as secondary outcome measures. We expect that it will take ~8 months to complete the study: 3 months for ethics review, 4 months to enroll 100 of a possible 200 eligible patients and 1 for data analysis.

This intervention will be judged primarily on its effect on length of stay for this population. It is our working hypothesis that this intervention will shorten length of stay by approximately 5 days. It will do this because TDCS will improve depression (GDS less than 5/15) and anxiety symptoms (score less than 9/30) and thus increase motivation and engagement. Readiness to proceed with therapy is a clinical judgement based on patient demeanour and GDS made by the Unit team who will be blind with respect to whether the patient is receiving TDCS or part of the sham group. Data will include: demographics: gender, age and diagnosis. Geriatric Anxiety Inventory, Geriatric Depression and Quality of Life scales will be completed within 1 week of admission, and at ~ 3 and 5 weeks (+3 days) after intervention initiated. Testing will be coordinated with the Unit Occupational Therapist to avoid duplication or the risk of over testing.

Data analysis:

1. Baseline group statistics (mean age &, standard deviation, male/female count, diagnostic frequencies, initial mean & standard deviations of GDS, Geriatric Anxiety Inventory and Quality of Life scores).
2. Effect of length of stay: Student t test will be used to determine if there is a significant difference between the 2 groups, defined as p<0.05.
3. Changes in Depression, anxiety or quality of life: significant differences from baseline at 3 and 5 weeks intervals will be assessed based on minimum clinical differences using a chi squared test.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 65 years old
* a Geriatric Depression Score above 4
* cognitively sound enough to give consent
* know English well enough to understand the procedure

Exclusion Criteria:

* being treated for an infection

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2020-02-09 (Actual)

PRIMARY OUTCOMES:
Length of stay | average length of stay varies from 28 to 42 days
  How long the patient is in hospital measured in days

SECONDARY OUTCOMES:
Geriatric Depression Score | applied within 1 week of admission and then at 3 and 5 weeks
  Survey assessing depression level of subject
Geriatric Anxiety Score | applied within 1 week of admission and then at 3 and 5 weeks
  Survey assessing anxiety level of subject
Older Person Quality of Life Questionnaire | applied within 1 week of admission and then at 3 and 5 weeks
  Survey assessing subject's impression of thier overall quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Kammerer, MD, Principal Investigator — Alberta Health services
Locations (1):
- Glenrose Rehabilitation Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We may also use the depression, anxiety and quality of life (QofL) results to look at the effects of direct current stimulation on symptoms of depression and anxiety.

REFERENCES:
- [Background] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Derived] Figeys M, Villarey S, Leung AWS, Raso J, Buchan S, Kammerer H, Rawani D, Kohls-Wiebe M, Kim ES. tDCS over the left prefrontal Cortex improves mental flexibility and inhibition in geriatric inpatients with symptoms of depression or anxiety: A pilot randomized controlled trial. Front Rehabil Sci. 2022 Oct 25;3:997531. doi: 10.3389/fresc.2022.997531. eCollection 2022. PMID 36386776
- See also: Adverse events of tDCS and tACS: A review. Hideyuki Matsumoto a,⇑, Yoshikazu Ugawa. Clinical Neurophysiology Practice 2 (2017) 19-25 — http://doi.org/10.1016/j.cnp.2016.12.003